CLINICAL TRIAL: NCT04544215
Title: A Clinical Study of Allogeneic Human Adipose-derived Mesenchymal Progenitor Cell Exosomes (haMPC-Exos) Nebulizer for the Treatment of Carbapenem-resistant Gram-negative Bacilli-induced Pulmonary Infection
Brief Title: A Clinical Study of Mesenchymal Progenitor Cell Exosomes Nebulizer for the Treatment of Pulmonary Infection
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic, patient enrollment was slower than expected. After enrolling 26 patients, the trial was suspended as our partner company stopped producing haMPC-Exos.
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEXDR
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-05

CONDITIONS: Drug-resistant
Keywords: human adipose-derived mesenchymal progenitor cell exosomes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MPCs-derived exosomes Dosage 1 (Experimental): low-dose group
  Interventions: Biological: Dosage 1 of MPCs-derived exosomes
- MPCs-derived exosomes Dosage 2 (Experimental): high-dose group
  Interventions: Biological: Dosage 2 of MPCs-derived exosomes
- No exosomes (Placebo Comparator): No MPCs-derived exosomes
  Interventions: Biological: No MPCs-derived exosomes

INTERVENTIONS:
Biological: Dosage 1 of MPCs-derived exosomes — 7 times aerosol inhalation of MPCs-derived exosomes (8.0*108 nano vesicles/3 ml at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7).
  Arms: MPCs-derived exosomes Dosage 1
Biological: Dosage 2 of MPCs-derived exosomes — 7 times aerosol inhalation of MPCs-derived exosomes (16.0*108 nano vesicles/3 ml at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7).
  Arms: MPCs-derived exosomes Dosage 2
Biological: No MPCs-derived exosomes — No aerosol inhalation of MPCs-derived exosomes
  Arms: No exosomes

SUMMARY:
Evaluate the efficacy and safety of haMPC-Exos treatment with pulmonary infection caused by gram-negative bacilli resistant to carbapenems.

DETAILED DESCRIPTION:
Pulmonary infection is a critical disease threatening human health. With the extensive use of antibiotics, the incidence of clinical drug resistance has been on the rise significantly in recent years. Once drug resistance occurs, we will see a high mortality rate due to scarce therapies and a poor prognosis. It is almost impossible to surmount the severe pulmonary infection caused by drug-resistant bacteria only by upgrading antibiotics. The commonly used supportive therapies clinically, such as glucocorticoids and immunomodulators, also lack forceful medical evidence. Therefore, it is urgent to explore new treatments.

Mesenchymal stem/progenitor cell exosomes are nano-sized vesicles secreted by mesenchymal stem/progenitor cells under certain conditions, which contain a lot of proteins, lipids and nucleic acids with tissue repair and immunomodulatory functions.

Mesenchymal stem/progenitor cell exosomes are nano-sized vesicles secreted by mesenchymal stem/progenitor cells under certain conditions, which contain a lot of proteins, lipids and nucleic acids with tissue repair and immunomodulatory functions.

Currently, it has been confirmed that stem cells can visibly improve the pathological changes of lungs caused by infection, lighten pulmonary edema, reduce protein exudation, mitigate alveolar inflammation, and remove bacteria. Thus, it brings new hope for the treatment of pulmonary infection caused by extensively drug-resistant bacteria.

Patients were treated, in the research project, with well-suited noninvasive haMPC-Exos aerosol inhalation, in an attempt to verify the efficacy and safety of haMPC-Exos treatment with pulmonary infection caused by gram-negative bacilli resistant to carbapenems.

ELIGIBILITY:
Inclusion Criteria:

- 1.Willingness of study participant to accept this treatment arm, and signed informed consent; 2.Male or female, aged at 18 years (including) to 75 years old; 3.Hospital-acquired pneumonia (HAP), including ventilator-associated pneumonia (VAP), was diagnosed within 48 h. The diagnosis must simultaneously comply with the three clinical and radiological criteria described below, which occurred more than 2 d (48 h) after hospitalization, within 7 d after discharge (HAP) or at least 2 d (48 h) after mechanical ventilation (VAP):

1. The patients had at least one of the following clinical manifestations:

   * New or deteriorating pulmonary symptoms or signs, such as cough, dyspnea, shortness of breath (e.g., respiratory rate higher than 25 beats/min), expectoration or need for mechanical ventilation;
   * Hypoxemia (e.g., when subjects breathe room air at standard atmospheric pressure, the partial pressure of oxygen measured as lower than 60 mmHg by arterial blood gas [ABG], or the ratio of partial pressure of oxygen to fraction of inspired oxygen [PaO2/FiO2] deteriorated);
   * According to the deterioration of oxygenation (ABG or PaO2/FiO2), the support system for the ventilator should be replaced urgently to strengthen oxygenation, or the positive end-expiratory pressure level should be changed;
   * Aspirable respiratory secretions newly appeared;
2. The patients had at least one of the following signs:

   * Confirmed fever (e.g., body temperature ≥ 38.4℃);
   * Hypothermia (e.g., body temperature ≤ 35℃);
   * Total peripheral white blood cell (WBC) count ≥ 11 × 109/L;
   * Leukopenia, and total WBC ≤ 4 × 109/L;
   * Immature neutrophils (rod-shaped nuclear cells) > 15% was observed on peripheral blood smears;
3. The chest X-ray of the patients showed new or progressive infiltration, and pneumonia was considered.

4.The pathogenic test of the lower respiratory tract specimens revealed carbapenem-resistant Gram-negative bacilli (Pseudomonas aeruginosa, Klebsiella pneumoniae or Acinetobacter baumannii), which were consistent with the drug resistance spectrum and intermediate or resistant to all carbapenem antibiotics, namely, the minimum inhibitory concentration (MIC) of meropenem or imipenem ≥ 2 μg/ml (2 μg/ml was intermediate and 4 μg/ml was drug-resistant). The MIC of ertapenem ≥ 1 μg/ml, of which 1 μg/ml was intermediate and ≥ 2 μg/ml was drug-resistant.

Exclusion Criteria:

* 1.Patients with severe allergic constitution or positive skin test result for test products; 2.Confirmed or suspected community acquired pneumonia (CAP)； 3.Confirmed or suspected pneumonia caused by mycoplasma, chlamydia, legionella, viruses, fungi or parasites; 4.HAP/VAP caused by obstruction, including lung cancer (or other malignant disease that causes lung obstruction) or other known obstructions; 5.Active immunosuppression, it is defined as receiving immunosuppressive drugs or under medical conditions associated with immunodeficiency. Including: 1) HIV (AIDS or CD4 < 200 cells/mm3); 2) received chemotherapy within 6 weeks before randomization; 3) immunosuppressive therapy, including maintenance glucocorticoid therapy (> 40 mg/day Prednisolone equivalent dose); 4) absolute neutrophil count < 500 mg/mm3; additional condition for inclusion: 1) Short-term (within one week) systemic (intravenous or oral) steroid therapy, using steroids for the treatment of skin disorders; 6.History of epilepsy and requirement for continuous anticonvulsant treatment or anticonvulsant treatment received within the last 3 years; 7.Undergoing hemodialysis or peritoneal dialysis; 8.Estimated or actual rate of creatinine clearance < 15 ml/min; 9.It is expected that any of the following drugs will be used during the study: Within 2 weeks before screening, or continuous use of valproic acid or divalproex sodium; 5-selective serotonin reuptake inhibitor, tricyclic antidepressant, 5-HT1 receptor agonist (triptans) or monoamine oxidase inhibitor; monoamine oxidase inhibitor (MAOIs) (or use of MAOIs within 2 weeks before screening) pethidine; buspirone; traditional Chinese medicine or herbal medicine; 10.Lung transplantation； 11.Bone marrow transplantation； 12.History of deep venous thrombosis or pulmonary embolism within the last 3 months; 13.Undergoing ECMO or high-frequency oscillatory ventilation support; 14.The estimated survival time <8 days; 15.HIV, viral hepatitis type B，viral hepatitis type C，or syphilis infection; 16.Period of pregnancy or lactation, or planned pregnancy within 6 months; 17.Incapable of understanding study protocol; 18.Any condition of unsuitable for the study determined by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measures: | Up to 8 days
  1.Clinical cure rate on the 8th d

SECONDARY OUTCOMES:
1.Bacterial clearance rate on the 8th d; | Up to 8 days
  Bacterial clearance rate on the 8th d
2.Mortality on the 28th and 90th d; | Up to 28-90 days
  Mortality on the 28th and 90th d
3.Recurrence rate after cure within 28 d; | Up to 28 days
  Recurrence rate after cure within 28 d
4.Secondary infection rate of other pathogenic bacteria after cure within 28 d; | Up to 28 days
  Secondary infection rate of other pathogenic bacteria after cure within 28 d
5.Duration of mechanical ventilation within 28 d; | Up to 28 days
  Duration of mechanical ventilation within 28 d
6.Length of ICU stay (d) within 28 d; | Up to 28 days
  Length of ICU stay (d) within 28 d
7.Incidence of adverse reactions at the end of treatment and 28 d after initial treatment. | Up to 28 days
  Incidence of adverse reactions at the end of treatment and 28 d after initial treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication